CLINICAL TRIAL: NCT01209858
Title: A Open-label Study to Investigate the Potential Pharmacokinetic Interaction of Perampanel With Oral Contraceptives in Healthy Female Subjects
Brief Title: A Study to Investigate the Potential Pharmacokinetic Interaction of Perampanel With Oral Contraceptives in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-E044-029
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Partial Onset Epilepsy
Keywords: epilepsy
MeSH Terms: conditions — Epilepsy | interventions — perampanel

ARMS (2):
- Experimental 1 (Experimental)
  Interventions: Drug: Perampanel and Microgynon-30
- Experimental 2 (Experimental)
  Interventions: Drug: Perampanel and Microgynon-30

INTERVENTIONS:
Drug: Perampanel and Microgynon-30 — Part A: Microgynon-30 single oral dose on Day 1 Period 1 and Day 35 Period 2; perampanel oral daily dose starting at 4 mg per day Period 2 from Days 1 through 35 and titrated weekly.
  Arms: Experimental 1
Drug: Perampanel and Microgynon-30 — Part B: Perampanel single oral dose of 6 mg on Day 1 Period 1 and Day 21 Period 2; Microgynon-30 orally from Day 1 through Day 21 of Period 2.
  Arms: Experimental 2

SUMMARY:
The purpose of this study is to investigate the effects of perampanel on the pharmacokinetics (PK) of a single-dose oral contraceptive (OC)containing ethinylestradiol (EE) and levonorgestrel (LN) (Microgynon-30) and to investigate the effects of repeated dosing of OC containing EE and LN (Microgynon-30) on the PK of a single dose of perampanel.

DETAILED DESCRIPTION:
This will be an open-label, non-randomized, fixed sequence study in healthy female subjects. The study has 2 parts: Part A investigating the effects of steady state perampanel on the pharmacokinetics (PK) of a single-dose oral contraceptive (OC) containing ethinylestradiol (EE) and levonorgestrel (LN) (Microgynon-30) and Part B investigating the effects of repeated dosing of an OC containing EE and LN (Microgynon-30) on the PK of a single dose of perampanel.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects, aged 18 - 55 years old inclusive at Screening;
2. Body mass index (BMI) within the range of 18-32 kg/m^2 inclusive at Screening;
3. Must not be taking any form of hormonal contraceptives, including hormonal intrauterine device (IUD), for at least 8 weeks prior to dosing;
4. All females must have a negative serum beta human chorionic gonadotropin (B- hCG) test result at Screening and negative urine B-hCG test result at each Baseline. Females of child-bearing potential must agree to use 2 medically acceptable methods of contraception (eg, abstinence where this is the subject's preferred lifestyle, a non-hormonal intrauterine device, a double-barrier method such as condom + spermicide or condom + diaphragm with spermicide, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 4 weeks after study drug discontinuation. The only subjects who will be exempt from this requirement are postmenopausal women (defined as at least 12 months consecutive amenorrhea, in the appropriate age group, without other known or suspected primary cause) or subjects who have been sterilized surgically or who are otherwise proven sterile (ie, bilateral tubal ligation with surgery at least 1 month prior to dosing, hysterectomy, or bilateral oophorectomy with surgery at least 1 month prior to dosing);
5. With no known contraindication to Microgynon-30;
6. Are willing and able to comply with all aspects of the protocol; and
7. Provide written informed consent.

Exclusion Criteria:

1. Have evidence of clinically significant cardiovascular, hepatic, gastrointestinal, renal, respiratory, endocrine, hematological, neurological, or psychiatric disease or abnormalities or a known history of any gastrointestinal surgery (including cholecystectomy) that could impact the PK of the study drug;
2. Have a known history of clinically significant drug or food allergies or are presently experiencing seasonal allergies;
3. Have an inability to tolerate venipuncture and/or venous access;
4. Have a history of alcohol abuse (within the past 6 months) or who drink more than the maximum recommended number of units of alcohol per week (14 units for women) or who are unwilling to abstain from consumption of alcohol throughout the periods of in-patient confinement;
5. Have a history of drug abuse or dependence or have a positive result from a urine drug screening test;
6. Received any experimental drug within the 12 weeks leading up to the start of study drug treatment or who are currently enrolled in another clinical trial;
7. Smoke more than 5 cigarettes (or equivalent amount of tobacco) per day or who are unwilling to abstain from the use of nicotine-containing products throughout the period of in-patient confinement;
8. Consume more than 5 caffeinated beverages per day (eg, 5 cups of tea, coffee or cans of cola) or who are unwilling to abstain from consumption of caffeine-containing food and beverages throughout the periods of in-patient confinement;
9. Have taken any inhibitor of CYP450 within 2 weeks prior to the first dosing (eg, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or Seville orange products);
10. Donated blood or blood products within 12 weeks prior to the start of dosing or who intent to donate blood during the study or within 8 weeks of completion of the study;
11. With a QTcF interval greater than 450 msec at Screening or either Baseline or a family history of prolonged QTc syndrome or sudden death;
12. With a positive result Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCVAb) screen at Screening;
13. Have been diagnosed with acquired immune deficiency syndrome (AIDS), or test positive for human immunodeficiency virus (HIV) at Screening;
14. With a positive alcohol test at Screening or at either Baseline;
15. With a Screening hemoglobin below the lower limit of normal [LLN] and/or with hematological parameters consistent with acute or chronic blood loss (hematocrit [Hct] below the LLN, mean corpuscular hemoglobin [MCH] below LLN and mean corpuscular hemoglobin concentration [MCHC] below LLN);
16. Taking, or have taken, any prescribed or over-the-counter drug or herbal remedies in the 2 weeks prior to Screening (unless the OTC drug has a long half-life [ie, 5 x t1/2 greater than 2 weeks]) with the exception of paracetamol, which is allowed up to 12 hours prior to dosing;
17. Within 4 weeks prior to dosing, are on special diets or have taken dietary aids that are known to induce CYP3A4 (eg, St John's Wort); or
18. Have a known personal or family history of arterial/venous thrombosis.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Part A: Pharmacokinetics (PK) of ethinylestradiol (EE) and levonorgestrel (LN) | Up to 24 hours postdose on Days 1 (Tr Pd 1) and 35 (Tr Pd 2).
Part B: Pharmacokinetics (PK) of perampanel | Up to 72 hours postdose on Days 1 (Tr Pd 1) and 21 (Tr Pd 2).

CONTACTS AND LOCATIONS:
Overall Officials: Prof Tim Mant, Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles Ltd, London, United Kingdom